CLINICAL TRIAL: NCT06728150
Title: Study Investigating the Role of Routine Screening and Molecular Characterisation of Brain Metastasis in the Management of High-risk Metastatic Breast Cancer
Acronym: STORM
Status: Not yet recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other); Breast Cancer Trials, Australia and New Zealand (Other)
Responsible Party: Principal Investigator, Mahesh Iddawela, Associate Professor, Monash University
Other Study IDs: Project 331/22
Record Dates: First submitted 2024-11-13; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Metastatic; Brain Metastasases
Keywords: Breast cancer brain metastases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissues form past breast cancer or brain metastases tissues and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: computerized tomography — The patients will have 3 monthly CT scans of the brain for 2 years and 6 monthly CT scans for 2 years for total of 4 years.

SUMMARY:
The purpose of this study is to improve outcome of breast cancer patients who develop brain metastases. This will investigate the benefits of early detection of brain metastases using brain imaging.

In patients diagnosed and currently being treated for advanced or metastatic breast cancer, current guidelines do not recommend routine brain imaging. However, there is emerging evidence suggesting that patients diagnosed without symptoms of brain metastases may have a better outcome than those with symptoms such as headache, vomiting and weakness.

In current practice, if signs and symptoms suggestive of brain metastases are to develop, then the doctor will arrange imaging of the brain, which may be a computerised tomography (CT scan) and/or a magnetic resonance imaging (MRI) scan. Should brain metastasis be detected, local radiotherapy, chemotherapy or targeted treatments will be offered.

When initially diagnosed with metastatic or advanced breast cancer, participant will or would have undergone a brain scan by either MRI or CT during normal standard full-body CT scan (chest, abdomen and pelvis) imaging. In this study, each time participants have a regular full-body CT scans to assess treatment progress, they will also have an additional CT scan of the brain.

Participants will have a total of 12 extra brain scans, with scans taking place every three months for the first 2 years, and every 6 months for the following years. These scans will occur at the same location as your current treatment. There will be no extra costs involved in the study and participants will be in the study for 4 years and following their follow-up details will be collected from medical records.

Some participants who develop brain metastases during the followup will have neurosurgery to remove these metastases. The investigators will collect either fresh or archived tissues and a cerebrospinal fluid (CSF) sample at the time of surgery from those patients.

If the treating investigators do not think neurosurgery is an option, they will ask participants to have a lumbar puncture for the collection of CSF. The purpose of this optional CSF collection is to take a liquid biopsy to check for markers (or biomarkers) potentially expressed by the breast cancer tumour cells in the brain. Participants will also be asked to provide a blood sample as well as old tumour from breast surgery (other metastatic tumour tissue).

The information obtained from this component of the study will not impact a parcipants current management, but it will help researchers to develop better treatments for breast cancer brain metastases in the future.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer with visceral, nodal or bone metastasis
* Human epidermal growth factor type2 (HER2-positive disease)
* Triple negative breast cancer (TNBC) with metastatic disease
* Oestrogen Receptor Positive disease (ER-positive disease) after second-line therapy and cyclin dependent kinase 4/6 inhibitors (CDK4/6 inhibitors), plus more than two sites of bone metastasis or visceral metastasis
* Diagnosis of metastatic disease in the last 3 months and free of symptoms or disease (with brain MRI confirmation) • Medicare Eligible

Exclusion Criteria:

* Symptomatic brain metastasis
* Inability to provide consent
* Inadequate organ function
* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with a diagnosis of metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of screen-detected asymptomatic brain metastasis. | 12 months
  CT scan of the brain used to determine evidence of new metastases.

SECONDARY OUTCOMES:
Incidence of symptomatic brain metastases | Though to study completion, an average of 1 year
  CT scans of the brain
Progression free survival | Though to study completion, an average of 1 year
  Time form entry into the study to brain metastases development
Overall survival | Though to study completion, an average of 1 year
  Time form entry into the study to death
Number of surgical resections | Though to study completion, an average of 1 year
  The number of patients who develop brain metastases having surgery
Rate of stereotactic radiotherapy | Though to study completion, an average of 1 year
  The number of patients having stereotactic radiotherapy assesses using medical records
Evaluation of the role of early treatment on intracranial disease control | Though to study completion, an average of 1 year
  Time form initial surgical or radiotherapy or observation to progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Iddawela, MBBS FRACP PhD, Principal Investigator — Associate Professor and Medical Oncologist
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The details of the protocol, patient information sheet, de-identified data and analysis
Supporting Information: Study Protocol
Time Frame: After 4 years
Access Criteria: With ethics approval from The Alfred ethics committee.